CLINICAL TRIAL: NCT01551615
Title: A Phase I, Open-label, Single-center Study to Assess the Pharmacokinetics of Metformin, an OCT2 Substrate, in Healthy Subjects When Administered Alone and in Combination With a Single Oral Dose of Vandetanib (CAPRELSA) 800 mg
Brief Title: A Phase I Study to Assess the Pharmacokinetics of Metformin When Administered Alone and in Combination With Vandetanib
Acronym: Vandetanib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D4200C00102
Record Dates: First submitted 2012-03-05; First posted 2012-03-13 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: Phase 1; healthy volunteers; pharmacokinetics; vandetanib; metformin; AUC(0-t); t1/2; tmax; CL/F; Vz/F; Cmax
MeSH Terms: interventions — Metformin; vandetanib

ARMS (1):
- Metformin then metformin + vandetanib (Experimental): Metformin alone followed by metformin in combination with vandetanib
  Interventions: Drug: Metformin 1000 mg; Drug: Vandetanib 800 mg

INTERVENTIONS:
Drug: Metformin 1000 mg — 2 x 500 mg oral tablets
Drug: Vandetanib 800 mg — 2 x 300 mg and 2 x 100 mg oral tablets

SUMMARY:
Study in Healthy Volunteers to Assess the Pharmacokinetics of Metformin Administered Alone and In Combination with Vandetanib

DETAILED DESCRIPTION:
A Phase I, Open-label, Single-center Study to Assess the Pharmacokinetics of Metformin, an OCT2 Substrate, in Healthy Subjects When administered Alone and in Combination with a Single Oral Dose of Vandetanib (CAPRELSA) 800 mg

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females aged 18 to 50 years with a weight of at least 50 kg and a body mass index between 18 and 30 kg/m2 inclusive.
* Females must have a negative pregnancy test at screening, must not be lactating and must be of non-childbearing potential.
* Volunteers will be wild type for the OCT2 gene (as tested for within the last 6 months prior to Day 1 in Period 1)

Exclusion Criteria:

* History or presence of gastrointestinal, hepatic, or renal disease or any medically significant disorder.
* History of or ongoing severe allergy/hypersensitivity to drugs with a similar chemical structure or class to vandetanib or metformin.
* Volunteers who smoke more than 5 cigarettes per day or are unable to refrain from smoking while resident in the study center.
* Known or suspected history of drug abuse.
* Screening supine blood pressure of greater than 140/90 mmHg and/or a resting heart rate of less than 45 beats per minute.
* Clinically significant current active skin disease (eg moderate to severe acne, psoriasis, eczema).
* Any positive result on screening for serum hepatitis B, surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
AUC for metformin administered alone and in combination with vandetanib 800 mg | Period 1: Predose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 32, 40, 48, 60, 72, and 96 hours post dose. Period 2: pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 32, 40, 48, 60, 72, and 96 hours post-dose.
Cmax for metformin administered alone and in combination with vandetanib 800 mg | Period 1: Predose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 32, 40, 48, 60, 72, and 96 hours post dose. Period 2: pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 32, 40, 48, 60, 72, and 96 hours post-dose.

SECONDARY OUTCOMES:
Frequency and severity of adverse events | Treatment period 7-14 days
ECG data | Treatment period 7-14 days
Laboratory data | Treatment period 7-14 days
Vital signs data | Treatment period 7-14 days
Other PK parameters for metformin administered alone and in combination with vandetanib 800 mg | Period 1: Predose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 32, 40, 48, 60, 72, and 96 hours post dose. Period 2: pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 32, 40, 48, 60, 72, and 96 hours post-dose.
Vandetanib PK parameters for vandetanib in combination with metformin | Period 2: pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 18, 24, 36, 48, 72, 96, 168, 240, 336, 504, and 672 hours post-dose.
PK parameters for metformin in urine when administered alone and in combination with vandetanib | Period 1: Day 1, 0 to 24 hrs and 24 to 48 hrs post metformin dose. Period 2: Day 1, 0 to 24 hrs and 24 to 48 hrs post metformin dose.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Johansson S, Read J, Oliver S, Steinberg M, Li Y, Lisbon E, Mathews D, Leese PT, Martin P. Pharmacokinetic evaluations of the co-administrations of vandetanib and metformin, digoxin, midazolam, omeprazole or ranitidine. Clin Pharmacokinet. 2014 Sep;53(9):837-47. doi: 10.1007/s40262-014-0161-2. PMID 25117183
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1437&filename=CSR-D4200C00102.pdf
- See also: CSR-D4200C00102.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1437&filename=CSR-D4200C00102.pdf
- See also: Revised_CSP_redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1437&filename=D4200C00102_Revised_CSP_redacted.pdf